CLINICAL TRIAL: NCT07023133
Title: Impact of Weight Loss on Mitochondrial Function
Acronym: WLMF
Status: Not yet recruiting | Type: Observational
Sponsor: Towson University (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Nicolas D. Knuth, Associate Professor, Towson University
Other Study IDs: 2340
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Weight Loss; Bariatric Surgery
Keywords: weight loss; bariatric surgery
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study cohort group: The study cohort will be made up of individuals that have self selected for bariatric surgery.
  Interventions: Behavioral: Weight loss

INTERVENTIONS:
Behavioral: Weight loss — All participants will have self selected for bariatric surgery and their weight loss and mitochondrial function will be measured in this study.

SUMMARY:
Loss of body weight can elicit an adaptive decline in energy expenditure during rest and physical activity beyond what is expected based on the loss of metabolically active tissue, a phenomenon termed metabolic adaptation. The weight loss-induced decrease in energy expenditure (i.e., altered energy efficiency) can hinder continued weight loss and contributes to variation in weight loss success. The molecular mechanisms responsible for metabolic adaption include changes to sympathetic nervous system activity, decreases in leptin and thyroid hormones, and increases in skeletal muscle mitochondrial efficiency and capacity, though the dominant mechanism for metabolic adaptation is unclear. We have recently shown, using near-infrared spectroscopy (NIRS) technology, that we can non-invasively assess skeletal muscle mitochondrial efficiency (i.e., oxygen consumption rate) and capacity. The purpose of this study is to evaluate the association between skeletal muscle mitochondrial efficiency and capacity after weight loss with metabolic adaption and weight loss variability. To accomplish this aim, we will recruit individuals with obesity who have elected for bariatric surgery at local bariatric centers. We will assess their energy expenditure and mitochondrial efficiency and capacity before and after weight loss.

DETAILED DESCRIPTION:
The procedures for this study involve two visit, one before bariatric surgery and one approximately 4 months after surgery, to our laboratory. The specific tests performed are listed below and are the same for each visit (each visit will take about 2 hours). Participants will be asked to arrive dressed in loose-fitting shorts that allow for assessments to be done on the lower leg.

Upon receipt of a signed consent form, a Demographics and Health History survey will be emailed to participants. Participants will be asked to complete the questionnaire in advance of their first in-person visit and will not be repeated at the second visit. The questionnaire will take ~10 minutes to complete and will be used to document any health conditions and medications.

Upon arrival for their in-person visit, we will measure the participant's seated blood pressure and heart rate as well as height and weight to calculate their body mass index (BMI). The following tests will then be performed:

1. Body Composition measurement: A DEXA scan will be performed while the participant lays on their back. A separate risk acknowledgment form for the DXA scan will be provided. Female participants of childbearing age who believe they may be pregnant or are not sure, will be offered a free pregnancy test prior to the DEXA scan.
2. Blood pressure (SphygmoCor) measurement: An automated pressure cuff will be placed on the participant's upper arm and inflated.
3. Resting whole-body metabolism. This assessment measures the amount of energy the body needs at rest (i.e., resting metabolic rate) to maintain normal bodily function and will take approximately 20 minutes. Participants will be asked to lie down and rest quietly while their expired breath, collected via an open hood worn over the head, will be analyzed for oxygen and carbon dioxide content to assess their resting metabolic rate.
4. Resting muscle metabolism: Muscle metabolism will be measured using near-infrared spectroscopy (NIRS), which is the typical use of the NIRS device. Specifically, a small mark will be placed on the center of the tibialis anterior (TA) muscle on the front of the dominant lower leg. An ultrasound machine will be used over the marked site on their muscle to capture an image and calculate the thickness of the TA muscle as well as the fat and skin layer over the muscle. Next, a small NIRS probe will be placed over the mark and secured into place with flexible wrap to minimize movement. There is no known risk associated with the NIRS device beyond potential irritation of the skin akin to the placement of any plastic device on the skin. NIRS measurements will be collected continuously through the duration of the test using blue-tooth. Small adhesive electrical stimulation pads will be placed on the TA muscle above and below the probe. A pneumatic blood pressure cuff will be placed around the thigh (upper leg) of their dominant leg just above the knee. The testing protocol will begin with resting measures that include 3 x 30s occlusions of the leg in which the blood pressure cuff will be inflated between 250-300mmHg. This will be followed by 30s stimulation of the muscle to mimic "exercise" to the TA muscle using electrical stimulation and then a series of short (6 x 5s) occlusions of the leg in which the blood pressure cuff will be again inflated between 250-300mmHg. The intensity of electrical stimulation is moderate and produces a tingling sensation and twitching of the muscle but is not painful. It provides a standardized muscle movement that mimics tapping of one's foot. This test will be repeated 4 times. When the repetitions are complete, the test will end with 5-minutes of blood pressure cuff occlusion and 3 minutes of data collection after the cuff is released.
5. Walking metabolism measurement: Participant's customary walking speed and metabolic cost (i.e. rate of oxygen consumption) will be measured at the level of the whole-body and at the level of the muscle during a 5-minute walking test performed over a 20-meter course. Distance traveled during the 5 minutes will be used to calculate their walking speed. Whole-body metabolic cost will be calculated from the measurement of oxygen consumption and carbon dioxide production rates while walking using a COSMED indirect calorimeter device. Specifically, participants will walk while wearing a facemask (for collection of expired breath) connected to the COSMED device harnessed to their back. The COSMED and harness weigh less than 3 pounds. Muscle oxygen consumption rate (i.e., metabolic cost) while walking will be measured using the NIRS device previously placed on the TA muscle. A pneumatic blood pressure cuff will be placed around the thigh (upper leg) of their dominant leg just above the knee and inflated between 250-300 mmHg for 10 seconds at the end of the walking to allow for measurement of muscle oxygen consumption rate during the occlusion. Participants will also wear a polar hear rate monitor around their chest for measurement of heart rate while walking; heart rate will be recorded by the COSMED device via Bluetooth. These measures are painless and non-invasive. Given that participants will walk at their normal, customary gait speed, no screening for any medical conditions will be used for exclusion beyond those listed above. There is no risk beyond that risk associated with normal ambulation given the self-selected walking speed.
6. Physical activity level. Objective daily physical activity data will be collected using a wrist-worn accelerometer. At the end of their visit, participants will be fitted with this watch-like device that is worn at the wrist, wear it for seven consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* obesity (BMI>30 kg/m2); self elected for bariatric surgery

Exclusion Criteria:

* body mass > 350 pounds; presence of type 2 diabetes, thyroid disease, coronary heart disease, congenital heart disease, peripheral arterial disease; having a pacemaker; the use of a walking aid; the presence of an injury that would modify normal gait; and women who are currently pregnant or trying to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with obesity that have self elected for bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 4 months
  The degree of weight loss after bariatric surgery
Mitochondrial function | 4 months
  Degree of change in mitochondrial function as a result of weight loss

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analyzed during the current study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: Beginning 1 year after publication with no end date.
Access Criteria: Access to study IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). Please contact corresponding author for more information or to submit a request.